CLINICAL TRIAL: NCT02122653
Title: Evaluation and Training of Muscle Fitness in Pre-frail Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung University (Other)
Responsible Party: Principal Investigator, Ya-Ju Chang, Professor, Chang Gung University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10044
Record Dates: First submitted 2014-04-23; First posted 2014-04-24 (Estimated); Last update posted 2014-04-24 (Estimated); Status verified 2014-04

CONDITIONS: Fatigue
Keywords: Fatigue; aging; transcranial magnetic stimulation; interpolated; twitch technique
MeSH Terms: conditions — Fatigue | interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Older WT (Experimental): Older people with weight training
  Interventions: Other: Weight training
- Older WT and ES (Experimental): Older people with weight training combined electrical stimulation.
  Interventions: Other: Weight training; Device: Electronic muscle stimulator
- Young control group (No Intervention): Young people with control group

INTERVENTIONS:
Other: Weight training — Participants will perform 4 weeks of Weight training for lower extremities.
  Arms: Older WT; Older WT and ES
Device: Electronic muscle stimulator — Participants will perform 4 weeks of electrical stimulation for Quadriceps muscle belly.
  Arms: Older WT and ES

SUMMARY:
Muscle strength and endurance are important indexes of fitness. The muscle strength is the most important single predict factor of functional ability in aged frail individuals. Frailty related muscle weakness and fatigue are adapted from the pre-frail stage. Finding the contributions of the central and the peripheral factors to the deficits of muscle fitness and developing an effective muscle fitness training program for pre-frail individuals are very important.

The muscle weakness and fatigue can be categorized into peripheral or central causes. The central fatigue and voluntary activation failure originate from the decrease in motivation or the reduction of the conduction within corticospinal tracts. Long term activation failure and central fatigue will cause disuse of muscle and result in peripheral weakness and peripheral fatigue. Studies found the selective type II fiber atrophy in aged people and this finding was different from the type I atrophy in conventional immobilization models. It is possible that the activation failure leads to the recruitment failure of high threshold type II fibers at the pre-frail stage. Quantifying the weighting of central versus peripheral factors contributing to the exercise limitation in pre-frail people is important.

Most of the conventional strength and endurance training programs are based on the researches of young groups. These programs are not able to prevent people become frail. It is possibly that, due to the limitation of central fatigue, the pre-frail individuals stop exercise before the effective intensity being achieved. Almost no training program has been design for enhancing the voluntary activation level and relief the central fatigue. Seeking an appropriate training program to enhance central activation at the pre-frail stage is very important for preventing people become frail.

Previous studies have shown that increasing afferent input by peripheral electrical stimulation (ES) at sensory threshold enhanced the plasticity of contralateral primary sensory cortex, the excitability of corticospinal tracts, and the functional performance in young adults. ES, which is easy to quantify the dose of afferent input, is a feasible method to be used in training. Combining afferent input with strength training might be able to overcome the central activation failure and help recruit high threshold motor unit in pre-frail individuals.

ELIGIBILITY:
Health subjects:

Exclusion Criteria:

Musculoskeletal injuries for knee. Osteoporosis. Diabetes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2012-08; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Muscle twitch force | Baseline, 4 weeks,8 weeks.
  Measure of changes in muscle twitch force by interpolation twitch technique.
Muscle voluntary activity level | Baseline, 4 weeks,8 weeks.
  Measure of changes in muscle voluntary activity level by interpolation twitch technique.
The central activation and the excitability of motor cortex | Baseline, 4 weeks,8 weeks.
  Measure of changes in the central activation and the excitability of motor cortex by Transcranial magnetic stimulation.
Muscle strength test for lower extremities. | Baseline, 4 weeks,8 weeks.
  Measure of changes in muscle strength test for lower extremities by clinical test.

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung University, Taoyuan District, Taiwan